CLINICAL TRIAL: NCT00005545
Title: Arterial Endothelial Function--An Epidemiologic Study
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Trudy L Burns, Professor, University of Iowa
Other Study IDs: 5088; R37HL061857 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Arteriosclerosis; Carotid Artery Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored plasma and DNA samples

SUMMARY:
To determine if risk factors measured in childhood can predict the development of atherosclerotic coronary and carotid artery disease in adulthood.

DETAILED DESCRIPTION:
BACKGROUND:

Many young adult subjects have some degree of atherosclerotic coronary and carotid artery disease and experience no symptoms. As time passes, many die suddenly and unexpectedly and only limited therapeutic process begins in youth, a measure of the early manifestations of atherosclerosis may have the potential of identifying subjects at risk for premature coronary and carotid occlusive vascular disease when therapeutic options can be administered. Impaired brachial artery flow mediated dilatory (FMD) capacities have been shown to exist in children and young adults with hypercholesterolemia, hyperhomocysteinemia, diabetes and in those who smoke. Impaired brachial artery FMD has been shown to related to impaired endothelial function, which is an early manifestation of the atherosclerotic process. If impaired brachial artery FMD is a predictor of the process, then it may be used to non-invasively assess atherosclerosis early in its development and to evaluate the effect of therapeutic interventions.

DESIGN NARRATIVE:

In this longitudinal study using previously studied members of the Muscatine study, measurements are made of contemporaneous risk factors, and brachial artery FMD, along with coronary artery calcification (CAC) and carotid artery intimal-medial thickness (IMT) (the latter two established measures of early atherosclerosis) and again three years later. The effort is designed to examine the following hypotheses: 1) Established risk factor levels measured in childhood, adulthood and across the years form childhood through adulthood are predictive of brachial artery flow mediated dilatory (FMD) capacities; 2) Putative risk factor levels measured in adulthood are related to the degree of brachial artery FMD, CAC and carotid artery IMT; 3) Brachial artery FMD, CAC and carotid artery IMTare related in adults; and 4) Brachial artery FMD is predictive of increased carotid artery IMT.

ELIGIBILITY:
Participated in at least on school survey examination, at least one young-adult follow-up survey examination and the first Longitudinal Adult Cohort examination

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Muscatine Study Longitudinal Adult Cohort - representative sample of childhood participants from the 1970s
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 1998-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation | 1999 to 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Lauer, Principal Investigator — University of Iowa

REFERENCES:
- [Background] Tschirren J, Lauer RM, Sonka M. Automated analysis of Doppler ultrasound velocity flow diagrams. IEEE Trans Med Imaging. 2001 Dec;20(12):1422-5. doi: 10.1109/42.974936. PMID 11811841